CLINICAL TRIAL: NCT05380765
Title: Developing a Positive Approach to Substance Use Prevention in North American Indian Adolescents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rhode Island (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: R34AA027619 (NIH)
Record Dates: First submitted 2022-04-22; First posted 2022-05-19 (Actual); Last update posted 2024-06-05 (Actual); Status verified 2024-06

CONDITIONS: Alcohol Drinking; Tobacco Use; Drug Use
MeSH Terms: conditions — Alcohol Drinking; Tobacco Use

STUDY DESIGN:
Intervention Model Description: wait-list control
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Native PATHS Condition (Experimental): A strengths-based, behavioral economic approach to increasing engagement and reinforcement for engaging in alternative activities.
  Interventions: Behavioral: Native PATHS
- Wait-List Control (No Intervention): Participants will receive the Native PATHS program once 6-month follow up surveys have been completed.

INTERVENTIONS:
Behavioral: Native PATHS — A strengths-based, behavioral economic approach to increasing engagement and reinforcement for engaging in alternative activities.
  Arms: Native PATHS Condition

SUMMARY:
The overall objective of this project is to develop and obtain preliminary data on acceptability, feasibility, and initial efficacy of Native PATHS. This work is guided by the stage model guidelines for treatment development and adaptation 25. Stage 1a will occur in two sequential steps. First, the investigators will recruit youth who are in 5th - 8th grade and their family members (N=24, 12 youth, 12 adults 18+) to participate in three talking circle sessions to obtain feedback on the cultural adaptation and implementation of the treatment. Next, the investigators will conduct an open label pilot (N=9). Youth and their family members, (up to 3 per youth) will provide qualitative and quantitative feedback after each session. In Stage 1b, 60 youth will participate in a pilot randomized controlled trial, testing the efficacy of the newly created program (n=30) against a wait list control (WLC) condition (n=30). Ultimately, this program of research is expected to result in a well-specified, efficacious prevention program that could be readily disseminated and generalizable to other Indigenous populations with minimal adaptation.

DETAILED DESCRIPTION:
Alcohol is one of the primary determinants of health disparity among many Indigenous populations with rates of alcohol-attributable mortality substantially higher than for Whites (73.8 per 100,000 vs. 27.5), and therefore, is a key threat to optimal health and well-being to Indigenous youth. Indigenous youth living in both the US and Canada tend to begin using alcohol, tobacco, and other drugs (ATOD) at earlier ages than most other ethnic/racial groups, and tend to move more quickly to regular use, resulting in earlier onset of ATOD disorders. Despite the severity of the problem, there continues to be an urgent unmet need for effective prevention programs that are culturally tailored to Indigenous populations of the US and Canada. The overall objective of this project is to develop and obtain preliminary data on the acceptability, feasibility, and initial efficacy of Native PATHS (Positive Approaches to reducing Harm from Substance Use). Native PATHS is a strengths-based, family prevention program for Indigenous youth in 5th-8th grade which focuses on delayed ATOD initiation. The development of Native PATHS has been guided by formative work in this community, taking a behavioral economic and positive psychological approach to prevention. Applied to prevention, behavioral economic theory focuses on reducing the availability of ATOD and increasing ATOD-free alternatives and the reinforcement received from engaging in ATOD-free activities. Activities in Native PATHS will work with families to help with establishing ATOD-free rules, limit physical availability of ATOD in the home, and reinforce youths' participation in ATOD-free activities. Positive psychological interventions (PPIs) focus on increasing positive emotions, life satisfaction, and well-being. PPIs will be used to enhance the enjoyment received from ATOD-free activities and to improve life satisfaction. Native PATHS is culturally consistent with North American Indigenous views of health that describe health in terms of a balance between the physical, spiritual, emotional, and mental aspects of life, which is represented in the teachings of the Medicine Wheel. Collaboratively, the investigators will work together with tribal partners on further adaptation of the program to include family and Indigenous ways of parenting in a culturally meaningful way. The overall goals proposed project will 1) finalize Native PATHS with participation from youth and family members in talking circles and an open pilot trial; 2) assess the effectiveness of Native PATHS in reducing ATOD initiation and intentions to use ATOD; 3) begin to evaluate the possible mechanisms/moderators of action including potential mediators future orientation and alternative reinforcer/activity engagement and reinforcement received, compared to a wait-list control group. The investigators will also evaluate positive affect as a potential moderator of any treatment effect, such that those higher in positive affect will be less likely to engage in ATOD use and be less likely to endorse intentions to use ATOD.

ELIGIBILITY:
Inclusion Criteria - Youth Participants:

1. residing in the First Nation community,
2. identify as a member of a First Nation,
3. be in grades 5th - 8th at time of enrollment, and
4. one youth per household may participate.

Inclusion Criteria - Family Participants:

1. at least 18 years of age
2. reside within the First Nation community
3. be identified, by the youth, as an important influence in their life
4. be committed to helping the youth make good decisions regarding using substances

Ages: 10 Years to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 60 (Estimated)
Dates: Start 2024-06-17 (Estimated); Primary Completion 2025-05-31 (Estimated); Study Completion 2025-05-31 (Estimated)

PRIMARY OUTCOMES:
Past month alcohol use | Baseline
  Respondents will be asked whether they have used alcohol in the past month (yes/no).
Past month alcohol use | End of treatment (up to 12 weeks following baseline)
  Respondents will be asked whether they have used alcohol in the past month (yes/no).
Past month alcohol use | Six months following end of treatment
  Respondents will be asked whether they have used alcohol in the past month (yes/no).
Past three-month alcohol use | Baseline
  Respondents will be asked whether they have used alcohol in the past three months (yes/no).
Past three-month alcohol use | End of treatment (up to 12 weeks following baseline)
  Respondents will be asked whether they have used alcohol in the past three months (yes/no).
Past three-month alcohol use | Six months following end of treatment
  Respondents will be asked whether they have used alcohol in the past three months (yes/no).
Past month marijuana use | Baseline
  Respondents will be asked whether they have used marijuana in the past month (yes/no).
Past month marijuana use | End of treatment (up to 12 weeks following baseline)
  Respondents will be asked whether they have used marijuana in the past month (yes/no).
Past month marijuana use | Six months following end of treatment
  Respondents will be asked whether they have used marijuana in the past month (yes/no).
Past three-month marijuana use | Baseline
  Respondents will be asked whether they have used marijuana in the past three months (yes/no).
Past three-month marijuana use | End of treatment (up to 12 weeks following baseline)
  Respondents will be asked whether they have used marijuana in the past three months (yes/no).
Past three-month marijuana use | Six months following end of treatment
  Respondents will be asked whether they have used marijuana in the past three months (yes/no).
Past month cigarette smoking | Baseline
  Respondents will be asked whether they have smoked cigarettes in the past month (yes/no).
Past month cigarette smoking | End of treatment (up to 12 weeks following baseline)
  Respondents will be asked whether they have smoked cigarettes in the past month (yes/no).
Past month cigarette smoking | Six months following end of treatment
  Respondents will be asked whether they have smoked cigarettes in the past month (yes/no).
Past three-month cigarette smoking | Baseline
  Respondents will be asked whether they have smoked cigarettes in the past three months (yes/no).
Past three-month cigarette smoking | End of treatment (up to 12 weeks following baseline)
  Respondents will be asked whether they have smoked cigarettes in the past three months (yes/no).
Past three-month cigarette smoking | Six months following end of treatment
  Respondents will be asked whether they have smoked cigarettes in the past three months (yes/no).
Alcohol use intentions | Baseline
  Respondent will be asked how often in the next month they think they will get drunk with friends and how often in the next month they would like to get drunk with friends, on a five-point scale from 0 (never) to 4 (10 or more times), where higher scores indicate more frequent intentions to use alcohol in the next month.
Alcohol use intentions | End of treatment (up to 12 weeks following baseline)
  Respondent will be asked how often in the next month they think they will get drunk with friends and how often in the next month they would like to get drunk with friends, on a five-point scale from 0 (never) to 4 (10 or more times), where higher scores indicate more frequent intentions to use alcohol in the next month.
Alcohol use intentions | Six months following end of treatment
  Respondent will be asked how often in the next month they think they will get drunk with friends and how often in the next month they would like to get drunk with friends, on a five-point scale from 0 (never) to 4 (10 or more times), where higher scores indicate more frequent intentions to use alcohol in the next month.
Cigarette smoking susceptibility | Baseline
  Cigarette smoking intentions will be measured using the Susceptibility to Smoking measure, which includes four items that asking respondents the likelihood that they will begin to smoke/experiment with cigarettes on a four-point scale from 0 (definitely not) to 3 (definitely yes), with higher scores indicating greater likelihood of intending to smoke cigarettes in the future.
Cigarette smoking susceptibility | End of treatment (up to 12 weeks following baseline)
  Cigarette smoking intentions will be measured using the Susceptibility to Smoking measure, which includes four items that asking respondents the likelihood that they will begin to smoke/experiment with cigarettes on a four-point scale from 0 (definitely not) to 3 (definitely yes), with higher scores indicating greater likelihood of intending to smoke cigarettes in the future.
Cigarette smoking susceptibility | Six months following end of treatment
  Cigarette smoking intentions will be measured using the Susceptibility to Smoking measure, which includes four items that asking respondents the likelihood that they will begin to smoke/experiment with cigarettes on a four-point scale from 0 (definitely not) to 3 (definitely yes), with higher scores indicating greater likelihood of intending to smoke cigarettes in the future.
Marijuana use intentions | Baseline
  Respondent will be asked how often in the next month they think they will use marijuana with friends and how often in the next month they would like to use marijuana with friends, on a five-point scale from 0 (never) to 4 (10 or more times), where higher scores indicate more frequent intentions to use marijuana in the next month.
Marijuana use intentions | End of treatment (up to 12 weeks following baseline)
  Respondent will be asked how often in the next month they think they will use marijuana with friends and how often in the next month they would like to use marijuana with friends, on a five-point scale from 0 (never) to 4 (10 or more times), where higher scores indicate more frequent intentions to use marijuana in the next month.
Marijuana use intentions | Six months following end of treatment
  Respondent will be asked how often in the next month they think they will use marijuana with friends and how often in the next month they would like to use marijuana with friends, on a five-point scale from 0 (never) to 4 (10 or more times), where higher scores indicate more frequent intentions to use marijuana in the next month.

CONTACTS AND LOCATIONS:
Overall Officials: Nichea S Spillane, Ph.D., Principal Investigator — University of Rhode Island
Locations (1):
- University of Rhode Island, Kingston, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: No